CLINICAL TRIAL: NCT03752320
Title: Usefulness of a Multiplex Polymerase Chain Reaction (mPCR) Assay for the Diagnosis of Postoperative Pneumonia After Thoracic Surgery
Brief Title: Multiplex Polymerase Chain Reaction in Postoperative Pneumonia After Thoracic Surgery
Acronym: POP-PCR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180010; 2018-A01908-47 (Other: ANSM)
Record Dates: First submitted 2018-08-30; First posted 2018-11-26 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Pneumonia; Bacterial Pneumonia
Keywords: Postoperative pneumonia; Thoracic surgery; Multiplex PCR; Bacterial and pulmonary colonization; Diagnosis; Mortality
MeSH Terms: conditions — Pneumonia; Pneumonia, Bacterial; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- POP+ and POP-: POP+: patients with postoperative pneumonia POP-: patients without postoperative pneumonia

SUMMARY:
Background: In thoracic surgery, postoperative pneumonia (POP) is the leading cause of postoperative morbidity and mortality. The clinical diagnosis of POP is difficult and conventional microbiological diagnostic tests perform poorly. The contribution of molecular diagnostic tests (multiplex PCR, mPCR) should be evaluated to optimize the diagnostic and therapeutic management of POP.

Objectives: The main objective is to describe the microbiological relationship between the existence of pre- (if available) and intra-operative bronchial and pulmonary bacterial colonization and the occurrence of POP. The secondary objectives are to analyze the contribution of the mPCR for the diagnosis of POP and to validate the predictive factors of POP described in the literature Material and methods: A monocentric prospective non-interventional research with minimal risks and constraints. The study population is represented by all the consecutive adult patients hospitalized for lung surgical resection (except surgical resection indicated for infectious disease) during one year. The preoperative respiratory samples within the 3 preceding months (date and type, pathogen and threshold) are recorded, if available. Intra-operative bronchial aspirate is performed for direct examination and culture (pathogen and threshold) and mPCR (PCR1). A mPCR is optionally performed on the surgical specimen (PCR2). In case of postoperative clinical suspicion of POP, invasive or non invasive samples of respiratory tract secretions are obtained for direct examination and culture (pathogen, threshold) and mPCR (PCR3). A clinical pulmonary infection score (CPIS) is calculated by integrating the results of conventional tests (CPIS1) and mPCR (CPIS2).

The pre / intra operative and postoperative microbiological relationship will be described qualitatively and quantitatively and analyzed using correlation tests. Concordances and discrepancies between conventional tests and mPCR will be studied to analyze the contribution of molecular tests in this context.

DETAILED DESCRIPTION:
Background: Post operative pneumonia (POP) is a common and severe complication associated with a high morbidity and mortality, regardless of the type of surgery. In thoracic surgery, the global incidence of POP is estimated at 25%. Pre-operative bronchial and pulmonary bacterial colonization appear as a major risk factor for the occurrence of POP, according to the literature.

The diagnosis of POP is challenging, because the usual diagnostic criteria are poorly relevant and clinical diagnostic scores are not validated, which may explain the scarcity of published data in the literature.

Patients' fragility and comorbid conditions mainly due to smoking limit the opportunity to perform invasive microbiological diagnostic tests, and those latter perform poorly. Altogether, the pathogen(s) involved are identified in 14% to 50%.

The evaluation of the diagnostic contribution of molecular diagnostic tests (mPCR) is important in this context. Molecular diagnostic tests offer better performance (sensitivity and sensibility) than conventional test, and the results are not affected by previous exposure to antibiotics. These tests could be useful to analyze the microbiological relationship between pre or per-operative bronchial and pulmonary colonization and postoperative infection, to optimize the diagnostic and the management of POP after thoracic surgery.

Materials and methods: In this study, The investigators aim to describe the microbiological relationship between the existence of pre- (if available) and intra-operative bronchial and pulmonary bacterial colonization and the occurrence of POP. The investigators also intend to analyze the contribution of mPCR for the diagnosis of POP.

For more precision, primary and secondary outcomes descriptions are fully detailed in the corresponding section.

The investigators perform a monocentric prospective non-interventional research with minimal risks and constraints. The study population is represented by all the consecutive adult patients hospitalized for lung surgical resection (except surgical resection indicated for infectious disease) during one year at Tenon Hospital, a University teaching hospital in Paris, France. About 200 patients per year undergo a lung surgical resection. Depending on the POP incidence, the number of patients suspected of POP may vary between 25 and 50 during the study period. Study duration participation corresponds to the hospital length of stay.

PCR Film Array Pneumonia is the molecular test used in this study. It is designed to detect the most common and critical pathogens of pneumonia (bacteria, virus). The results are reported quantitatively. Patients' management is in line with recommendations and not modified by the research. The expected risks are those of the usual care.

The practical progress of the study is defined by:

* Preoperative. Patients' clinical characteristics, respiratory status and expected surgery data are collected. The preoperative respiratory samples (date and type, pathogen and threshold) are recorded if available within the 3 preceding months
* Per-operative. Intra-operative bronchial aspirate is performed for direct examination and culture (pathogen and threshold) and mPCR (PCR1). Surgery characteristics are collected. Per-operative antibioprophylaxis is in line with recommendations.
* Post operative. Identification of post operative complications (respiratory and extra respiratory) including POP. POP diagnosis is based on clinical and microbiological data (Clinical Pulmonary Infection Score). In case of clinical suspicion of POP, respiratory samples are performed for direct examination and culture (pathogen and threshold) and mPCR (PCR2). A CPIS score is calculated with conventional microbiological tests results (CPIS 1) and PCR results (CPIS2). Hospital health care and vital status at discharge are recorded.

Primary and secondary outcomes measures are fully detailed in the corresponding section.

Statistical analysis: The statistical analysis will be performed at the end of the study. The characteristics of the patients will be described and compared between two groups, i.e. patients with POP and patients without POP. Qualitative variables will be described by size and frequency, and quantitative variables by mean and standard deviation or median and inter-quartile range. Between-groups comparisons will be performed using a Chi2 or a Fisher exact test for qualitative variables, and a Student t test or Mann-Whitney U test for the quantitative variables.

For the primary outcome, the proportion of patients for whom the intra operative colonization strain and the postoperative infection strain are the same will be calculated (with their 95% confidence interval).

For the secondary outcomes, the overall concordance rate, and the qualitative and quantitative diagnostic discrepancies will be calculated with their 95% confidence interval between conventional and molecular tests. The proportions of patients with appropriate antibiotic therapy and with targeted antibiotic therapy will be estimated and compared between conventional and molecular tests.

The predictive factors for POP occurrence will be assessed by a logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients hospitalized for lung surgical resection
* Consenting to research

Exclusion Criteria:

* surgical resection indicated for infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the consecutive adult patients hospitalized for lung surgical resection (except surgical resection indicated for infectious disease) for one year at Tenon hospital, a University teaching in Paris, Assistance publique - Hôpitaux de Paris, France.
  About 200-250 patients undergo a thoracic surgery per year and are supported in the thoracic surgery department of Tenon hospital. If we consider a 25% incidence rate of post operative pneumonia, we expect 50-60 patients to be included during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients in whom the preoperative microorganism (colonization) is the same than that identified in POP. | Defined by the patient's hospitalization, from surgery to hospital discharge, until 28 days of follow up
  The diagnosis of POP is based on the CPIS using clinical data and microbiology (CPIS1 and CPIS2).
  The final diagnosis is:
  Certain: Clinical evidence of pneumonia, quantitative positive respiratory tract samples (RTS) above the thresholds Probable: Strong clinical suspicion (CPIS>6), RTS below the thresholds, no ongoing or recently introduced antibiotics (atb); or RTS below the thresholds with ongoing or recently introduced atb, regardless the clinical suspicion Possible: Low clinical suspicion (CPIS≤6), RTS below the thresholds, no ongoing or recently introduced atb; or CPIS≤6, negative RTS and ongoing or recently introduced atb Unlikely: Negative RTS with no ongoing or recently introduced atb; or CPIS≤6, negative RTS and ongoing or recently introduced atb.
  Comparing CPIS1 and CPIS2, we also asses the diagnostic contribution of molecular tests

SECONDARY OUTCOMES:
The rate of diagnostic concordance between conventional and molecular tests in the context of post operative pneumonia in thoracic surgery. | Defined by the patient's hospitalization, from surgery to hospital discharge, including the period management of post operative pneumonia, until 28 days of follow up
  Conventional and mPCR tests concordance is defined by the identification of the same microbiological species above or below the thresholds positivity for both tests.
  Qualitatively minor discrepancy is defined by different microbiological species below the thresholds for both tests.
  Qualitatively major discrepancy is defined by different microbiological species with both tests and below the threshold for one and above for the other.
  Quantitatively minor discrepancy is defined by the identification of the same microbiological species with both tests but below the positivity threshold for one and above for the other.
  Quantitatively major discrepancy is defined by the identification of different microbiological species above the thresholds for both tests.
Mesure of the theoretical impact of molecular diagnostic test results on the antibiotics use. | Defined by the patients' hospitalization, from surgery to hospital discharge, including the period management of post operative pneumonia, until 28 days of follow up
  A panel of independent clinicians will suggest a fictive antibiotic therapy based on mPCR results.
  The proportions of patients with appropriate antibiotic therapy and patients with targeted antibiotic therapy will be compared, according to the results of the microbiological tests (conventional vs. mPCR) for the initial empirical antibiotic therapy, and the secondary antibiotic therapy (at 24 and 48h).
The measurement of the association of general characteristics, pneumological and functional respiratory characteristics related to the surgical procedure with the occurrence of POPs in the entire study population. | Defined by the patient's hospitalization, from surgery to hospital discharge, including the period management of post operative pneumonia, until 28 days of follow up
  The predictive factors of post operative pneumonia described in the literature General, lung functional and surgical characteristics of patients will be recorded at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Martoukh, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Réanimation et USC médico-chirurgicale Hôpital Tenon, AP-HP, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No
individual participant data collected in this study will be used for publication.